CLINICAL TRIAL: NCT03781011
Title: Investigation on Clinical Application of Oral Carnitine Challenge Test as a Guidance of Personalized Nutrition for Patients With Cardiovascular Disease
Brief Title: Oral Carnitine Challenge Test Guides Personalized Nutrition for CV Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201712030RIND
Record Dates: First submitted 2018-12-10; First posted 2018-12-19 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2020-10

CONDITIONS: Dietary Modification; Cardiovascular Diseases
Keywords: Gut microbiota; Trimethylamine N-oxide; Oral carnitine challenge test; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants identified as high-TMAO producers through the oral carnitine challenge test will be invited to participate in a two-month vegetarian diet intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vegetarian diet intervention (Experimental): Patients identified as high-TMAO producers through the oral carnitine challenge test will be invited to participate in a two-month vegetarian diet intervention, supervised by a registered dietitian.
  Interventions: Behavioral: Vegetarian diet intervention

INTERVENTIONS:
Behavioral: Vegetarian diet intervention — Patients will received dietary education and supervision by dietician to avoid high carnitine/choline foods including red meat, eggs...etc.

SUMMARY:
The investigators plan to use the recently developed oral carnitine challenge test (OCCT) as a tool to exam individual's trimethylamine N-oxide (TMAO) production capacity from their gut microbiota. By using data collected by OCCT, the investigators defined subjects as high-TMAO producer or low-TMAO producer and apply low carnitine/choline diet as dietary intervention for the high-TMAO producers. After dietary intervention for two months, the investigators conducted OCCT for the participants and compare the TMAO production capacity before and after the dietary intervention.

DETAILED DESCRIPTION:
Patients diagnosed with cardiovascular disease at the CV clinics are being recruited to undergo the Oral Carnitine Challenge Test (OCCT) to assess the TMAO production capacity of their gut microbiota. Participants identified as high-TMAO producers will be invited to partake in a two-month vegetarian diet intervention, supervised by a registered dietitian, followed by a three-month period of reverting to their regular diet. The OCCT will be conducted before and after the vegetarian diet intervention, as well as after the diet recovery phase. Fecal samples will be collected and analyzed at the baseline, in the second month, and in the fifth month of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with risks of cardiovascular disease (CAD) or CAD patients proved by coronary angiography

Exclusion Criteria:

* age < 20, hx of GI surgery, hx of malignancy, antibiotic or probiotic or carnitine supplement use within one month, liver cirrhosis, end stage chronic renal disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
TMAO production capacity | Baseline, at the second month (following a two-month vegetarian diet intervention), and at the fifth month (after resuming a regular diet for three months).
  TMAO production capacity is measured by calculating the area under the curve of TMAO levels (quantification by LC-MS/MS) during the procedure of oral carnitine challenge test

SECONDARY OUTCOMES:
Compositional and functional changes of gut microbiota | Baseline, at the second month (following a two-month vegetarian diet intervention), and at the fifth month (after resuming a regular diet for three months).
  The compositional and functional changes of gut microbiota will be evaluated by shotgun metagenome sequencing. Taxonomy will be calculated as relative abundance of species-level genome bins (SGBs) and specific bacteria genes will be quantified as Reads Per Kilobase per Million (RPKM).

CONTACTS AND LOCATIONS:
Overall Officials: Ming-shiang Wu, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan